CLINICAL TRIAL: NCT01152645
Title: Phase II Study of ARQ 197 Monotherapy for Previously Treated Advanced/Recurrent Gastric Cancer
Brief Title: Study of ARQ 197 Monotherapy
Acronym: ARQ 197-004
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Kyowa Kirin Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ARQ 197-004
Record Dates: First submitted 2010-06-25; First posted 2010-06-29 (Estimated); Last update posted 2017-03-15 (Actual); Status verified 2017-03

CONDITIONS: Gastric Cancer
Keywords: Advanced/recurrent gastric cancer
MeSH Terms: conditions — Stomach Neoplasms | interventions — ARQ 197

ARMS (1):
- ARQ 197 (Experimental)
  Interventions: Drug: ARQ 197

INTERVENTIONS:
Drug: ARQ 197 — Orally twice daily administration of ARQ 197

SUMMARY:
A phase II open-label study with ARQ 197 administered orally and twice daily as monotherapy in patients with previously treated advanced/recurrent gastric cancer. The primary endpoint is disease control and the secondary efficacy endpoints include antitumor effect (tumor response), progression-free survival and overall survival. The pharmacokinetic profile and the safety profile are also evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Japanese or Korean with voluntary written informed consent for study participation
* A histologically or cytologically confirmed advanced/recurrent gastric cancer
* One or two prior chemotherapy regimens for advanced/recurrent gastric cancer
* At least one measurable lesion
* ECOG performance status of 0 or 1
* Life expectancy ≥3 months

Exclusion Criteria:

* Surgery for cancer within 4 weeks prior to the first dose of ARQ 197
* Confirmed other tumors than gastric cancer within 5 years prior to the first dose of ARQ 197
* Anticancer chemotherapy, hormone therapy, radiotherapy or immunotherapy within 2 weeks prior to the first dose of ARQ 197
* Positive for HIV antibody
* Known symptomatic brain metastasis
* Gastrointestinal disorders that could interfere with the absorption of ARQ 197 or operation history for gastrointestinal disorders
* Uncontrolled concomitant disease
* Patients who wish to have a child and who would not agree to use contraceptive measures
* Pregnant or lactating

Ages: 20 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2010-06; Primary Completion 2011-08 (Actual); Study Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
Antitumor effect | Tumor size was measured at Baseline, Day 29 and 54, and then every 6 week until discontinuation criteria met.
  Disease control

SECONDARY OUTCOMES:
Antitumor effect | Tumor size was measured at Baseline, Day 29 and 54, and then every 6 week until discontinuation criteria met.
  Tumor response
Progression-free survival | Tumor size was measured at Baseline, Day 29 and 54, and then every 6 week until discontinuation criteria met. In addition, survival was confirmed by biweekly inquiry during the study, and by follow up survey.
Overall survival | Survival was confirmed by biweekly inquiry during the study, and by follow up survey.
Pharmacokinetic profile | Plasma sample correction at pre-dose, 1, 2, 4, 6, 10, 12 and 24 hours on Day 1, and in addition, at pre-dose of Day 15 and 29.
  Plasma ARQ 197 concentrations and pharmacokinetic parameters following the first dose of ARQ 197
Adverse events | Patients will be monitored for occurrence of adverse events from the day of the first dosing to the completion of the examinations at the discontinuation of the study.

CONTACTS AND LOCATIONS:
Locations (2):
- Nagoya, Japan
- Seoul, South Korea